CLINICAL TRIAL: NCT02201953
Title: A Phase 3, Multicenter, Randomized, Open-Label Study to Compare the Efficacy and Safety of Sofosbuvir/GS-5816 Fixed Dose Combination for 12 Weeks With Sofosbuvir and Ribavirin for 24 Weeks in Subjects With Chronic Genotype 3 HCV Infection
Brief Title: Comparison of Sofosbuvir/Velpatasvir Fixed Dose Combination for 12 Weeks With Sofosbuvir and Ribavirin for 24 Weeks in Adults With Chronic Genotype 3 HCV Infection
Acronym: ASTRAL-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-1140; 2014-001682-27 (EudraCT Number)
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2016-09

CONDITIONS: Hepatitis C Virus Infection
Keywords: Sofosbuvir; Velpatasvir; SOF/VEL; GS-5816; Hepatitis C; HCV; Cirrhosis; Genotype 3
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — sofosbuvir-velpatasvir drug combination; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOF/VEL 12 Weeks (Experimental): SOF/VEL FDC for 12 weeks
  Interventions: Drug: SOF/VEL
- SOF+RBV 24 Weeks (Experimental): SOF+RBV for 24 weeks
  Interventions: Drug: SOF; Drug: RBV

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg FDC tablet administered orally once daily
  Other Names: Epclusa®; GS-7977/GS-5816
  Arms: SOF/VEL 12 Weeks
Drug: SOF — 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
  Arms: SOF+RBV 24 Weeks
Drug: RBV — Tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: SOF+RBV 24 Weeks

SUMMARY:
The primary objectives of this study are to compare the efficacy of treatment with sofosbuvir/velpatasvir (SOF/VEL) fixed-dose combination (FDC) for 12 weeks with that of sofosbuvir (SOF) + ribavirin (RBV) for 24 weeks and to evaluate the safety and tolerability of each treatment regimen in participants with chronic genotype 3 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV RNA ≥ 10^4 IU/mL
* HCV genotype 3
* Chronic HCV infection (≥ 6 months)
* Females of childbearing potential must have a negative serum pregnancy test
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception

Exclusion Criteria:

* Current or prior history of clinically-significant illness (other than HCV) that may interfere with subject treatment, assessment or compliance with the protocol
* Screening ECG with clinically significant abnormalities
* Laboratory results outside of acceptable ranges at Screening
* Pregnant or nursing female or male with pregnant female partner
* Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson's disease, alfa-1 antitrypsin deficiency, cholangitis)
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2014-07; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McNally, PhD, Study Director — Gilead Sciences
Locations (69):
- United States (24):
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - Aurora, Colorado
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Wellington, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lutherville, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - New York, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Germantown, Tennessee
  - San Antonio, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
- Australia (8):
  - Darlinghurst, New South Wales
  - Brisbane, Queensland
  - Clayton, Victoria
  - Fitzroy, Melbourne, Victoria
  - Melbourne, Victoria
  - Fremantle, Western Australia
  - Perth, Western Australia
  - Camperdown
- Canada (6):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Montreal, Quebec
  - Toronto
- France (11):
  - Clermont-Ferrand
  - Clichy
  - Créteil
  - Lille
  - Limoges
  - Lyon
  - Marseille
  - Paris
  - Pessac
  - Toulouse
  - Villejuif
- Germany (8):
  - Frankfurt am Main, Hessin
  - Cologne, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Hufelandstr, North Rhine-Westphalia
  - Berlin
  - Hamburg
  - Hanover
  - München
- Italy (2):
  - San Giovanni Rotondo, Foggia
  - Florence
- New Zealand (2):
  - Auckland
  - Christchurch
- San Juan, Puerto Rico
- United Kingdom (7):
  - Plymouth, Devon
  - Portsmouth, Hampshire
  - Glasgow
  - London
  - Manchester
  - Nottingham
  - Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Asselah T, Charlton M, Feld J, Foster GR, Mcnally J, Brainard DM, et al. The ASTRAL Studies: Evaluation of SOF/GS-5816 Single Tablet Regimen for the Treatment of Genotype 1-6 HCV Infection [Poster P1332]. J Hepatol 2015;62:S855-S6.
- [Result] Mangia, A., Roberts, SK., Pianko, S., Thompson, A at al. Sofosbuvir/GS-5816 Fixed Dose Combination for 12 Weeks Compared to Sofosbuvir with Ribavirin for 24 Weeks in Genotype 3 HCV Infected Patients: The Randomized Controlled Phase 3 ASTRAL-3 Study. Hepatology 2015; 62: 1 (SUPPL) 338A.
- [Result] Foster GR, Afdhal N, Roberts SK, Brau N, Gane EJ, Pianko S, Lawitz E, Thompson A, Shiffman ML, Cooper C, Towner WJ, Conway B, Ruane P, Bourliere M, Asselah T, Berg T, Zeuzem S, Rosenberg W, Agarwal K, Stedman CA, Mo H, Dvory-Sobol H, Han L, Wang J, McNally J, Osinusi A, Brainard DM, McHutchison JG, Mazzotta F, Tran TT, Gordon SC, Patel K, Reau N, Mangia A, Sulkowski M; ASTRAL-2 Investigators; ASTRAL-3 Investigators. Sofosbuvir and Velpatasvir for HCV Genotype 2 and 3 Infection. N Engl J Med. 2015 Dec 31;373(27):2608-17. doi: 10.1056/NEJMoa1512612. Epub 2015 Nov 17. PMID 26575258
- [Derived] Jacobson IM, Bourgeois S, Mathurin P, Thuluvath P, Ryder SD, Gerken G, Hernandez C, Vanstraelen K, Scherbakovsky S, Osinusi A, Tedesco D, Foster GR. The tolerability of sofosbuvir/velpatasvir for 12 weeks in patients treated in the ASTRAL 1, 2 and 3 studies: A pooled safety analysis. J Viral Hepat. 2023 May;30(5):448-454. doi: 10.1111/jvh.13814. Epub 2023 Mar 2. PMID 36740893
- [Derived] Younossi ZM, Stepanova M, Feld J, Zeuzem S, Sulkowski M, Foster GR, Mangia A, Charlton M, O'Leary JG, Curry MP, Nader F, Henry L, Hunt S. Sofosbuvir and Velpatasvir Combination Improves Patient-reported Outcomes for Patients With HCV Infection, Without or With Compensated or Decompensated Cirrhosis. Clin Gastroenterol Hepatol. 2017 Mar;15(3):421-430.e6. doi: 10.1016/j.cgh.2016.10.037. Epub 2016 Nov 12. PMID 27847279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, North America, Europe, and New Zealand. The first participant was screened on 14 July 2014. The last study visit occurred on 15 December 2015.
Pre-assignment Details: 652 participants were screened.
Groups:
- SOF/VEL 12 Weeks: Sofosbuvir/velpatasvir (SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet administered orally once daily for 12 weeks
- SOF+RBV 24 Weeks: Sofosbuvir (SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) administered orally for 24 weeks
Period: Overall Study
Arm/Group | SOF/VEL 12 Weeks | SOF+RBV 24 Weeks
Started | 278 | 280
Completed | 258 | 224
Not Completed | 20 | 56
Not completed — Randomized but Never Treated | 1 | 5
Not completed — Lack of Efficacy | 9 | 30
Not completed — Lost to Follow-up | 8 | 8
Not completed — Withdrew Consent | 2 | 5
Not completed — Adverse Event | 0 | 5
Not completed — Death | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug.
Groups:
- SOF/VEL 12 Weeks: SOF/VEL (400/100 mg) FDC tablet administered orally once daily for 12 weeks
- SOF+RBV 24 Weeks: SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) administered orally for 24 weeks
- Total: Total of all reporting groups
Arm/Group | SOF/VEL 12 Weeks | SOF+RBV 24 Weeks | Total
Number analyzed (Participants) | 277 | 275 | 552
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10.4) | 50 (10.0) | 50 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 101 | 208
  Male | 170 | 174 | 344
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 266 | 263 | 529
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 3 | 1 | 4
  White | 250 | 239 | 489
  Asian | 23 | 29 | 52
  American Indian or Alaska Native | 1 | 3 | 4
  Native Hawaiian or Pacific Islander | 0 | 2 | 2
  Not Disclosed | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  New Zealand | 9 | 8 | 17
  Canada | 15 | 18 | 33
  United States | 60 | 60 | 120
  Italy | 7 | 11 | 18
  United Kingdom | 58 | 47 | 105
  Australia | 49 | 44 | 93
  France | 48 | 52 | 100
  Germany | 31 | 35 | 66
HCV Genotype [Number; unit: participants]
  Genotype 3 (No Confirmed Subtype) | 9 | 18 | 27
  Genotype 3a | 265 | 250 | 515
  Genotype 3b | 2 | 5 | 7
  Genotype 3h | 0 | 2 | 2
  Genotype 3k | 1 | 0 | 1
Cirrhosis Status [Number; unit: participants]
  Yes | 80 | 83 | 163
  No | 197 | 187 | 384
  Missing | 0 | 5 | 5
IL28b Status [Number; unit: participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 105 | 111 | 216
    CT | 148 | 133 | 281
    TT | 24 | 31 | 55
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2 (0.72) | 6.3 (0.71) | 6.3 (0.72)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 86 | 81 | 167
  ≥ 800,000 IU/mL | 191 | 194 | 385
Prior HCV Treatment Experience [Number; unit: participants]
  Treatment-Naive | 206 | 204 | 410
  Treatment-Experienced | 71 | 71 | 142

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks | SOF+RBV 24 Weeks
Number analyzed (Participants) | 277 | 275
percentage of participants | 95.3 [92.1 to 97.5] | 80.7 [75.6 to 85.2]
Statistical Analysis 1: Comparison: SOF/VEL 12 Weeks vs SOF+RBV 24 Weeks; Test type: Non-Inferiority or Equivalence — Primary analyses consisted of non-inferiority test of Group 1 (SOF/VEL 12 weeks) versus Group 2 (SOF+RBV 24 weeks) at the 0.05 significance level. Non-inferiority was assessed using the conventional confidence interval approach and a non-inferiority margin of 10% was applied. The two-sided 95% confidence intervals was constructed using stratum-adjusted Mantel-Haenszel proportions, stratified by the randomization stratification factors (i.e cirrhosis status and prior treatment experience); Difference in proportions = 14.4, 95% CI 2-sided [9.2 to 19.6] — Difference in proportions between treatment groups and associated 95% confidence intervals (CI) are calculated based on stratum-adjusted Mantel-Haenszel proportions
Statistical Analysis 2: Comparison: SOF/VEL 12 Weeks vs SOF+RBV 24 Weeks; If the lower bound of 95% CI on the difference was > -10%, the p-value tested for the superiority of SOF/VEL for 12 weeks over SOF+RBV for 24 weeks. Superiority was demonstrated if the two-sided p-value is less than 0.05; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — P-value was from the Cochran-Mantel-Haenszel test stratified by cirrhosis status and prior HCV treatment experience

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks | SOF+RBV 24 Weeks
Number analyzed (Participants) | 277 | 275
percentage of participants | 0 | 3.3

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 are defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks | SOF+RBV 24 Weeks
Number analyzed (Participants) | 277 | 275
percentage of participants
  SVR4 | 96.8 [93.9 to 98.5] | 82.2 [77.1 to 86.5]
  SVR24 | 95.3 [92.1 to 97.5] | 80.7 [75.6 to 85.2]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Weeks 1, 2, 4, 6, 8, 10, 12, 16, 20, and 24
Time Frame: Weeks 1, 2, 4, 6, 8, 10, 12, 16, 20, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks | SOF+RBV 24 Weeks
Number analyzed (Participants) | 277 | 275
percentage of participants
  Week 1 (SOF/VEL: N = 277; SOF+RBV: N = 275) | 18.4 [14.0 to 23.5] | 17.5 [13.2 to 22.5]
  Week 2 (SOF/VEL: N = 276; SOF+RBV: N = 274) | 62.0 [55.9 to 67.7] | 50.0 [43.9 to 56.1]
  Week 4 (SOF/VEL: N = 276; SOF+RBV: N = 272) | 91.7 [87.8 to 94.6] | 88.2 [83.8 to 91.8]
  Week 6 (SOF/VEL: N = 276; SOF+RBV: N = 269) | 96.7 [93.9 to 98.5] | 98.9 [96.8 to 99.8]
  Week 8 (SOF/VEL: N = 276; SOF+RBV: N = 269) | 99.6 [98.0 to 100.0] | 99.3 [97.3 to 99.9]
  Week 10 (SOF/VEL: N = 276; SOF+RBV: N = 268) | 100.0 [98.7 to 100.0] | 99.3 [97.3 to 99.9]
  Week 12 (SOF/VEL: N = 275; SOF+RBV: N = 265) | 100.0 [98.7 to 100.0] | 99.6 [97.9 to 100.0]
  Week 16 (SOF/VEL: N = 0; SOF+RBV: N = 262) | NA [NA to NA] — Participants in the SOF/VEL group were only treated for 12 weeks. | 98.9 [96.7 to 99.8]
  Week 20 (SOF/VEL: N = 0; SOF+RBV: N = 260) | NA [NA to NA] — Participants in the SOF/VEL group were only treated for 12 weeks. | 99.6 [97.9 to 100.0]
  Week 24 (SOF/VEL: N = 0; SOF+RBV: N = 255) | NA [NA to NA] — Participants in the SOF/VEL group were only treated for 12 weeks. | 100.0 [98.6 to 100.0]

5. Secondary Outcome: Change From Baseline in HCV RNA at Weeks 1, 2, 4, 6, 8, 10, 12, 16, 20, and 24
Time Frame: Baseline; Weeks 1, 2, 4, 6, 8, 10, 12, 16, 20, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL 12 Weeks | SOF+RBV 24 Weeks
Number analyzed (Participants) | 277 | 275
log10 IU/mL
  Change at Wk 1 (SOF/VEL: N =272; SOF+RBV: N =268) | -4.26 (0.644) | -4.16 (0.640)
  Change at Wk 2 (SOF/VEL: N =274; SOF+RBV: N =272) | -4.82 (0.769) | -4.79 (0.702)
  Change at Wk 4 (SOF/VEL: N =276; SOF+RBV: N =270) | -5.02 (0.776) | -5.09 (0.699)
  Change at Wk 6 (SOF/VEL: N =275; SOF+RBV: N =269) | -5.06 (0.718) | -5.13 (0.712)
  Change at Wk 8 (SOF/VEL: N =276; SOF+RBV: N =269) | -5.07 (0.728) | -5.13 (0.712)
  Change at Wk 10 (SOF/VEL: N =276; SOF+RBV: N =267) | -5.07 (0.723) | -5.14 (0.710)
  Change at Wk 12 (SOF/VEL: N =275; SOF+RBV: N =264) | -5.08 (0.721) | -5.14 (0.711)
  Change at Wk 16 (SOF/VEL: N = 0; SOF+RBV: N = 262) | NA (NA) — Participants in the SOF/VEL group were only treated for 12 weeks. | -5.11 (0.765)
  Change at Wk 20 (SOF/VEL: N = 0; SOF+RBV: N = 259) | NA (NA) — Participants in the SOF/VEL group were only treated for 12 weeks. | -5.14 (0.715)
  Change at Wk 24 (SOF/VEL: N = 0; SOF+RBV: N = 255) | NA (NA) — Participants in the SOF/VEL group were only treated for 12 weeks. | -5.14 (0.715)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL 12 Weeks | SOF+RBV 24 Weeks
Number analyzed (Participants) | 277 | 275
percentage of participants | 4.0 | 14.2

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Groups:
- SOF+RBV 24 Weeks: SOF 400 mg tablet once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 24 weeks
Arm/Group | SOF/VEL 12 Weeks | SOF+RBV 24 Weeks
Serious Adverse Events (participants affected / at risk) | 6/277 | 15/275
Other Adverse Events (participants affected / at risk) | 216/277 | 243/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL 12 Weeks (N=277) | SOF+RBV 24 Weeks (N=275)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Propionibacterium infection (Infections and infestations) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Ruptured cerebral aneurysm (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL 12 Weeks (N=277) | SOF+RBV 24 Weeks (N=275)
Anaemia (Blood and lymphatic system disorders) | 1 | 25
Abdominal pain (Gastrointestinal disorders) | 10 | 19
Constipation (Gastrointestinal disorders) | 13 | 21
Diarrhoea (Gastrointestinal disorders) | 20 | 21
Dyspepsia (Gastrointestinal disorders) | 9 | 30
Nausea (Gastrointestinal disorders) | 47 | 58
Vomiting (Gastrointestinal disorders) | 8 | 20
Asthenia (General disorders) | 16 | 26
Fatigue (General disorders) | 71 | 105
Pyrexia (General disorders) | 4 | 14
Bronchitis (Infections and infestations) | 6 | 14
Nasopharyngitis (Infections and infestations) | 34 | 33
Decreased appetite (Metabolism and nutrition disorders) | 8 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 20
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 15
Disturbance in attention (Nervous system disorders) | 7 | 14
Dizziness (Nervous system disorders) | 15 | 21
Headache (Nervous system disorders) | 90 | 90
Anxiety (Psychiatric disorders) | 7 | 21
Insomnia (Psychiatric disorders) | 32 | 74
Irritability (Psychiatric disorders) | 23 | 40
Sleep disorder (Psychiatric disorders) | 9 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 22
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 20
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 25
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 35
Rash (Skin and subcutaneous tissue disorders) | 15 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years